CLINICAL TRIAL: NCT00985634
Title: Randomized Clinical Evaluation of LeGoo™ Internal Vessel Occluder Vs Traditional Vessel Loops
Brief Title: Clinical Evaluation of LeGoo™ Internal Vessel Occluder Versus Traditional Vessel Loops
Acronym: LeGoo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pluromed, Inc. (Industry)
Responsible Party: James Wilkie / Vice President Operations, Pluromed, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LeGoo EURO rev D
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Off Pump Coronary Artery Bypass Surgery
Keywords: off pump bypass OPCAB; OPCAB

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LeGoo (Experimental): Subjects in this arm, which is assigned at random, will receive the study device.
  Interventions: Device: LeGoo
- Control (Active Comparator): Subjects in this arm will not receive the study device, but receive the standard of care for vessel occlusion (vessel loops.)
  Interventions: Device: Control

INTERVENTIONS:
Device: LeGoo — LeGoo internal vessel occluder. Usage (dose) as required and determined by surgeon.
  Arms: LeGoo
Device: Control — Vessel loops
  Arms: Control

SUMMARY:
The primary purpose of this study is to demonstrate the clinical safety and efficacy of LeGoo™ in comparison to a standard vessel occlusion method (i.e. vessel loops). Although LeGoo™ is suitable for use in any vascular surgery where temporary vessel occlusion is desired, this study specifically focuses on the use of LeGoo™ in off-pump coronary bypass (OPCAB), as a most sensitive model of adverse changes that may occur at any vascular site.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical efficacy of LeGoo™ as compared to a traditional vessel loop. LeGoo is a device that is intended to be used during surgical procedures to temporarily occlude blood vessels while forming an anastomosis. LeGoo™ will be evaluated in subjects undergoing off-pump coronary artery by-pass (OPCAB) surgery. This is a prospective, randomized trial with a 30-day follow-up period. Half of the eligible patients will be randomized to the experimental group (LeGoo™); and the other half to the control group (standard vessel loops).

LeGoo™ is polymer-based device which is comprised of a non-toxic and biocompatible gel that exists as a liquid at low temperatures and rapidly transitions to a solid at body temperature, forming a plug that can occlude blood vessels. LeGoo™ is injected into a blood vessel that is intended to be occluded, where it stays in a "plug" form for several minutes allowing the surgeon to work in a bloodless field. The gel dissolves with time (spontaneously) or can be reversed back to liquid instantly by cooling the site with ice or irrigating with cold saline. Once dissolved below a minimum concentration, the polymer can never re-solidify.

The primary research hypothesis is that surgeons will obtain a bloodless surgical field and achieve satisfactory hemostasis in a larger proportion of anastomoses using LeGoo™ than using a conventional temporary hemostasis technique.

Satisfactory hemostasis is defined by the surgeon who will quantitate his/her observation about the quality of the surgical field using the following scoring system:

1. - Excellent hemostasis (no bleeding)
2. - Minimal bleeding (bleeding does not interfere with suturing)
3. - Modest bleeding (required intermittent use of another device to control bleeding at the site of the anastomosis)
4. - Copious bleeding (required continuous use of another device)

"Excellent hemostasis" and "minimal bleeding" are considered "satisfactory hemostasis." Satisfactory hemostasis will constitute a treatment success for the purpose of evaluating the primary efficacy of LeGoo. The primary endpoint is the proportion of anastomoses in which satisfactory hemostasis is achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects undergoing elective off pump coronary artery bypass (OPCAB) surgery where the surgeon prospectively plans to use a vascular occlusion device.
2. >70% proximal stenosis of at least one target coronary artery, other than left main
3. Age: between the ages 18 -79 years
4. Gender: male and female
5. Subject is willing and able to participate in a clinical research study and provides informed consent.
6. Subject is able and willing to participate in required follow-up procedures.

Exclusion Criteria:

1. Previous cardiac surgery.
2. Left ventricular dysfunction (EF <40%)
3. >50% of left main coronary artery stenosis
4. Subjects with a logistic EuroScore equal to or greater than 10% as calculated by the euroscore.org calculator
5. Emergent Surgery: Subjects undergoing surgery before the start of the next working day following catheterization
6. Creatinine > 200 µmol/L
7. Bilirubin > 21 µmol/L
8. Subjects with chronic pulmonary disease [ FEV1 < 45% ]
9. Any subject who is deemed by the investigator, for any reason, not suitable or able to participate in a clinical research study.
10. Pregnant women. Women of childbearing age will require a pregnancy test within 10 days of the operation and will be excluded if the result is positive.
11. Women who are lactating.
12. Subjects who have undergone other investigational therapy within 30 days prior to the operation or who are scheduled to receive investigational therapy within six months of the operation.
13. Subjects suspected to have one intra-myocardial artery among the coronary arteries to be bypassed during that surgery.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The primary research hypothesis is that surgeons will obtain a bloodless surgical field and achieve satisfactory hemostasis in a larger proportion of anastomoses using LeGoo™ than using a conventional temporary hemostasis technique. | in operating room

SECONDARY OUTCOMES:
Total duration of the anastomosis, blood loss during the surgery, Time required to occlude the vessel, the number of units of blood transfused during hospitalization. | in operating room (day of surgery)
Safety will be measured by comparing a composite of four serious adverse events experienced by the treated and control groups: death, graft occlusion, myocardial damage, and low post procedure cardiac output. | one month post op

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik fur Herzchirurgie Herzzentrum Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Wimmer-Greinecker G, Bouchot O, Verhoye JP, Perrault LP, Borgermann J, Diegeler A, Van Garsse L, Rastan AJ. Randomized clinical trial comparing a thermosensitive polymer (LeGoo) with conventional vessel loops for temporary coronary artery occlusion during off-pump coronary artery bypass surgery. Ann Thorac Surg. 2011 Dec;92(6):2177-83. doi: 10.1016/j.athoracsur.2011.07.003. PMID 22115228